CLINICAL TRIAL: NCT06669000
Title: Time Required to Dissolve Urate Deposits in Patients with Gout
Brief Title: Time Required to Dissolve Urate Deposits
Acronym: ReViGoRe 40
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); ART VIGGO Association for Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP240644; 2024-A00937-40 (Other: IDRCB)
Record Dates: First submitted 2024-09-23; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-09

CONDITIONS: Gout
Keywords: Gout; Flares; Tophi; Urate levels; Urate deposits; Ultrasound; Allopurinol; Febuxostat
MeSH Terms: conditions — Gout | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Month 0 and Month 24: 1 EDTA tube 10 ml; 1 EDTA tube 5 ml; 1 Paxgen 2 ml Month 6 and Month 36: 1 EDTA tube 10 ml; 1 Paxgen 2 ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Gout patients treated according to a Treat-to-Dissolve strategy: Patients initiated with ULT (urate target less than 40 mg/L), and followed every 6 months with Ultrasound until complete urate dissolution
  Interventions: Diagnostic Test: Standard X-Rays; Diagnostic Test: Ultrasound; Diagnostic Test: DECT of feet; Biological: DNA sample; Biological: Serum collection

INTERVENTIONS:
Diagnostic Test: Standard X-Rays — - Standard X-Rays: feet (Month 0)
Diagnostic Test: Ultrasound — - Ultrasound (score 0-24): assessment for DC (Double Contour) sign (0-3), aggregates (0-3), tophi (0-3) at MTP1s (first metatarsophalangeal joints) and DC sign (0-3) at both knees, according to the OMERACT, every 6 months until complete dissolution of urate deposits.
Diagnostic Test: DECT of feet — DECT of feet: in tophaceous patients only (Month 0, Month 24)
Biological: DNA sample — DNA will be collected at Month 0
Biological: Serum collection — - Serum will be collected at Month 0, Month 6, Month 12, Month 18, Month 24 , Month 36 and Month 48. For OMICs and epigenetic studies: Month 0, Month 6, Month 24 and Month 36.

SUMMARY:
Gout is characterized by episodes of acute arthritis of the lower limbs due to intermittent activation of innate immunity in the joints where urate crystals have formed. These crystals occur when serum urate (SUA) levels have been above 70 mg/L for many years. They can be dissolved by lowering SUA levels to at least 60 mg/L (treat-to-target - T2T - strategy). Once the crystals are dissolved, patients are no longer symptomatic and are considered to be in remission (treat-to-dissolve - T2D - strategy).

The presence of crystals and their dissolution during treatment can be monitored by repeated ultrasound (US) scans of the feet and knees.

The time required for complete dissolution varies from patient to patient. ReViGore40 is a cohort designed to i) determine the time to complete dissolution of urate deposits in joints when SUA levels are maintained below 40 mg/L, ii) determine the factors (clinical, biological, genetic) associated with the time required for complete dissolution of urate deposits within joints.

DETAILED DESCRIPTION:
Patients with newly diagnosed gout according to the 2015 ACR/Eular criteria, not treated with urate-lowering therapy and with US evidence of urate deposition (feet, knees; ultrasound score ≥ 2/24) will be enrolled in the ReViGore40 cohort.

In all patients, SUA levels will be lowered with allopurinol or febuxostat (XOI) depending on renal function (eGFR greater or less than 30 ml/mn/m2) or uricosurics, by starting medications at a low dose and subsequent titration. The target SUA levels is less than 40 mg/L in all patients.

Patients will then be monitored by US every 6 months until complete urate crystals dissolution. An ultrasound score (min 0- max 24; 0 meaning no urate deposits and 24 the highest value for quantifying the extent of deposits) will be calculated for each US scan. Dissolution is considered to have been achieved when a score of 0/24 is reached on two successive US scans performed 6 months apart.

The Predictive Factors (clinical, biological, genetic) associated with the complete dissolution of urate deposits will be determined.

DECT (feet) will be performed only in tophaceous patients at M0 and M24. Each patient will receive a capillary urate point of care device for self-urate measurement. Patients will be contacted monthly by nurses for the first 6 months to ensure treatment compliance and SUA target attainment.

Blood samples will be collected at M0, M6, M24 and M36 for omic and epigenetic studies. Clinical data will be collected at M0, M6, M12, M24, M36 and M48. Change in Protein, Epigenetic and omic profils will be determined.

DNA for genetic studies will be collected at M0. Co-morbidities, particularly cardiovascular and hepatic, will be assessed at M6: coronary artery calcium (CAC) scoring and liver fibroscan.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Gout according to the ACR/Eular 2015 criteria
* SUA levels greater than 60 mg/L
* US score (MTP1s, knees) ≥2/24
* Informed consent Dated and signed voluntarily

Exclusion Criteria:

* Ongoing urate lowering therapy
* Severe and uncontrolled diseases such as cancer, cardiovascular or neurovegetative diseases
* Pregnant or breast-feeding women
* No affiliation to the French National Social Security System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gout patient managed according to a T2T (treat to target) strategy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Time required for complete dissolution of urate deposits | Change between baseline (month 0) and up to 48 months after initiation of ULT
  For each patient, urate deposit dissolution will be monitored by repeated US scans.
  The US features which will be recorded according to the Outcome Measures in Rheumatology (OMERACT) scoring system:
  * at MTP1s: the DC sign, tophi and aggregates
  * at the knees (femoral condyles): the DC sign. The aggregates will only be scored if the DC sign and/or tophus are present and if the aggregates are not located inside a tophus. For each site, the US features will be graded as follows: absent (0) possible (1) moderate (2) important (3). Thus, a score (0-24) will be calculated for each patient. A score of 0 means that there are no longer urate deposits, while a score of 24 means that there are a lot of urate deposits. Dissolution is considered to have been achieved when a score of 0/24 is reached on two successive US scans performed 6 months apart

SECONDARY OUTCOMES:
Number of flares | At Month 0, Month 6, Month 12, Month 18, Month 24, Month 30, Month 36, Month 48
  Flares is defined when 3 of the following 4 criteria are present:
  * Patient-defined flare
  * Pain at rest greater than 3 on a 0-10 point numerical rating scale.
  * Presence of at least one swollen joint.
  * Presence of at least one hot joint.
Health status as assessed by the EQ-5D-3L questionnaire | At Month 0, Month 6, Month 12, Month 24, Month 36, Month 48
  Health status as assessed by the EQ-5D-3L descriptive system comprising the following five dimensions:
  * Mobility,
  * Self-care,
  * Usual activities,
  * Pain/discomfort
  * Anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the most appropriate box. This decision results into a 1-digit number. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Patient self-rated health on a vertical visual analogue scale (EQ VAS) | At Month 0, Month 6, Month 12, Month 24, Month 36, Month 48
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale from 0 to 100, with 100 being the best health and 0 corresponding to the worst health.
Health status as assessed by the HAQ-ID questionnaire | At Month 0, Month 6, Month 12, Month 24, Month 36, Month 48
  The questionnaire includes 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities, with 4 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section.
  The 8 scores of the 8 sections are summed and divided by 8. The score obtained ranges from 0 to 3. The higher the score, the worse the state of health.
Proteins profils | Month 0, Month 6, Month 24, Month 36
  Change in plasma Proteins concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- APHP, Lariboisière Hospital, Rheumatology departement, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided